CLINICAL TRIAL: NCT00901862
Title: Magnetic Therapy in Migraine Prophylaxis; Placebo-Controlled, Double-Blind, Crossed Study
Brief Title: Magnetic Therapy in Migraine Prophylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: DANIEL SAN JUAN ORTA, Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 105/06
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Migraine
Keywords: Migraine; therapy; magnetic therapy; prophylaxis; prevention
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Active PEFs (Active Comparator): The pulsed electromagnetic fields were directed to the wrist. The model used has the form of a bracelet called Quantum MH-2MR which uses, as a source of power, an alkaline battery of 1.5 volts connected to an electronic circuit formed by two hybrid circuits of magnetic oscillation and a control system of all the generating frequency system.
  Interventions: Device: Pulsed magnetic fields (Quantum MH-2MR bracelet)
- 2 Sham (Sham Comparator): The sham machines were identical to the machines in actual operation in both phases of the study. The only difference was that the hybrid circuits crucial for the generation of the electromagnetic field had been removed.
  Interventions: Device: Sham pulsed magnetic fields (Quantum MH-2MR bracelet)

INTERVENTIONS:
Device: Pulsed magnetic fields (Quantum MH-2MR bracelet) — Pulsed magnetic fields
  Arms: 1 Active PEFs
Device: Sham pulsed magnetic fields (Quantum MH-2MR bracelet) — Hybrid circuits crucial for the generation of the electromagnetic field had been removed.
  Arms: 2 Sham

SUMMARY:
Background: The therapy with pulsed electromagnetic fields (PEFs) has been used as a therapeutic modality for at least 40 years. However, their effect in the migraine prophylaxis is unclear.

Objectives: Evaluate the prophylactic effectiveness of the therapy with PEFs in the handling of migraines.

Methodology: Placebo-controlled, randomized, double-blind, crossed clinical study.

DETAILED DESCRIPTION:
Migraine is a disease which considerably affects the individual, the family and society.[1-3] In spite of the recent advances in the symptomatic and preventive treatment of migraine, the relative effectiveness of many commonly used prophylactic medicines is not well established. Most of these drugs have indirect effects that force their suspension or their restriction of prescription to patients with certain pathologies. This fact reduces their clinic effectiveness. [4]

The therapy with pulsed electromagnetic fields (PEF's) has been used as a therapeutic modality for at least 40 years. One of its well acknowledged uses is the healing of non-union fractures, [5] although there are other medical conditions that have also been susceptible to be treated with this type of therapies, like migraine [6], Parkinson disease, [7] and epilepsia, [8] among others. Nevertheless, only a few published studies demonstrate the effectiveness of the PEF's in the handling of migraine. These studies have been carried out in a small number of patients, without control groups6 or for very short periods of time [6, 9] as to demonstrate a suitable prophylactic effect. Therefore, this placebo-controlled, double-blind, crossed clinical study was carried out in order to evaluate the prophylactic effectiveness of the therapy with PEF's in the handling of migraine.

METHODOLOGY

Patients:

The subjects were selected from the Clinic of Headache of our hospital from 2006 to 2007. All the patients included in the study aged between 18-55yrs and fulfilled the diagnose criteria of migraine with and without aura in agreement to the International Headache Classification, 2004. The study was conducted in accordance with Good Clinical Practice guidelines and the Declaration of Helsinki (1996). The protocol and statement of informed consent were approved by the Institutional Review Board. All the patients accepted to participate voluntarily and signed an informed consent. Patients with cluster, medicines overuse, post-traumatic headache, sinusitis or other headache types, women who were pregnant, became pregnant during the study or were lactating, patients who were under other prophylactic treatments of migraine or did not signed the informed consent were excluded from this study. Patients were allowed to continue with the medication for the acute attacks of migraine; which consisted of administering 30 mg of sublingual ketorolac every eight hours, in case of migraine. The investigator was supplied with a sealed code for each individual patient that would be opened in case of an emergency that required knowledge of the treatment being taken.

Study design:

This was a double-blind, randomized, placebo-controlled and crossed trial. Participants who satisfied the inclusion criteria entered a four week baseline run-in period to verify the frequency and intensity of attacks, followed by 3 months of the treatment with PEF's or placebo, and then a 1 week of wash-out period between treatments, and then crossover.

Evaluation of the activity of the Cephalea:

Subjects were provided with a diary to record frequency, duration and intensity of their attacks, as well as the use of the analgesic during the whole study period. The intensity of the pain was evaluated with the analogous scale of pain, which has shown to be highly profitable and effective. The pain was stratified in a scale from zero (no pain) to ten (the most intense pain that the subject has undergone by at least one second). The diaries used were the typical ones, which have shown a high effectiveness and that only require an entrance per migraine. The patients were classified as responders if one month after having received any of the therapies, they had a reduction equal or greater to 50% in the frequency of episodes of migraine.

Randomization and follow up:

The sociodemographic characteristics and the patterns of basal activity of the cephaleas were determined for all the patients. The 19 patients who fulfilled the inclusion criteria were allocated to treatment according to a computer generated randomization procedure with 4 consecutive balanced blocks of two patients (one active, one placebo). They were randomized, in a simple way, in two groups of exposition: the real and the placebo one. Patients were evaluated by the researchers at the third and sixth months of treatment. Along this time, the patients registered in their diaries the frequency and clinical characteristics of the episodes of cephaleas during both treatments.

Exposition to the PFEs or Placebo:

The PEF's were directed to the wrist. The model used has the form of a bracelet called Quantum MH-2MR which uses, as source of power, an alkaline battery of 1.5 volts connected to an electronic circuit formed by two hybrid circuits of magnetic oscillation and a control system of all the generating frequency system. The power of the variable magnetic field generated by the equipment varied from 0.64 to 1.4 Gaussian, whereas the spectrum generated by the main fixed frequencies went from 0 to 240 Hertz, the semi-fixed one went from 241 to 360 Hertz and the random one went from 361 to 170 Megahertz. The control system continuously ordered the fixed generation of magnetic signals with a frequency that differed in 0.1 Hertz to each other in the region of the spectrum between 0 and 240 Hertz. It also ordered the semi-fixed generation (a fixed and a random portion) of frequencies between 241 and 360 Hertz, as well as the random generation (only when the external presence of these frequencies was detected) of a frequency between 261 and 170 MHz.

The machines were set under verification of their functionality with a voltmeter every three months and any moment in case they had been exposed to water. This was carried out by an engineer who did not have contact with patients and who did not participate in their clinical evaluation or follow up. The participants could not feel if the machine was working and neither could they mention in which group they were. The machines of placebo were identical to the machines in actual operation in both phases of the study. The only difference was that the hybrid circuits crucial for the generation of the electromagnetic field had been removed. As the subjects could not feel the change, there was no possibility that the subjects had knowledge about which of the machines provided therapy and which ones did not. At any moment the researchers were blinded to distinguish which of the devices was active and which one was not. The patients carried the devices continuously, except when there was the risk of contaminating them with water, as when bathing.

Outcome measures:

The primary outcome measure was change from baseline in the number and peak severity of migraine attacks during each double-blind phase. The secondary outcome was the proportion of patients who responded to each treatment with at least a 50% reduction in migraine attacks relative to baseline. Safety was assessed by reports of adverse events.

Statistical analysis:

We used descriptive statistical, means and standard deviations. All statistical calculations were performed using a computer with the software SPSS version 13.0 for Windows

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-55 years
* Fulfilled the diagnose criteria of migraine with and without aura in agreement to the International Headache Classification, 2004

Exclusion Criteria:

* Patients with cluster, medicines overuse, post-traumatic headache, sinusitis or other headache types
* Women who were pregnant, became pregnant during the study or were lactating
* Patients who were under other prophylactic treatments of migraine or did not signed the informed consent were excluded from this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was change from baseline in the number and peak severity of migraine attacks during each double-blind phase | 3 months

SECONDARY OUTCOMES:
The secondary outcome was the proportion of patients who responded to each treatment with at least a 50% reduction in migraine attacks relative to baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: DANIEL SAN JUAN ORTA, MD, Principal Investigator — Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suárez
Locations (1):
- Instituto Nacional de Neurologia y Neurocirugía Manuel Velasco Suarez, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] San-Juan D, Pon AA, Pohls FZ, Del Castillo-Calcaneo Jde D, Perez-Neri I, Rios C. Peripheral pulsed electromagnetic fields may reduce the placebo effect in migraine patients that do not respond to the sham intervention in a randomized, placebo-controlled, double-blind, cross-over clinical trial. Complement Ther Med. 2012 Feb-Apr;20(1-2):31-7. doi: 10.1016/j.ctim.2011.09.006. Epub 2011 Oct 15. PMID 22305246